CLINICAL TRIAL: NCT03765242
Title: Retrospective Medical Chart Review Study for Atrial Fibrillation Patents Treated With Oral Anticoagulant
Brief Title: Evaluation of Safety and Effectiveness on Oral Anticoagulants
Acronym: RCR-OAC
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-698
Record Dates: First submitted 2018-11-26; First posted 2018-12-05 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient initiating warfarin
  Interventions: Other: Non-Interventional
- Patient initiating apixaban
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This study is to compare the risk of major bleeding among oral anticoagulant (OAC)-naïve non-valvular atrial fibrillation (NVAF) patients initiating treatment

ELIGIBILITY:
Inclusion Criteria:

* Individuals greater than or equal to 20 years old as of the index date
* At least 1 diagnosis of NVAF prior to or on index date, identified by any medical records
* Newly treated with warfarin or apixaban between 01-Jan-2011 to 31-Dec-2016. The first warfarin or apixaban prescription date during the identification period will be designated as the index date

Exclusion Criteria:

* Patient's medical records indicating pregnancy during the follow-up period
* Patient's medical records indicating taking warfarin, apixaban, dabigatran, rivaroxaban, or edoxaban during the 6-months prior to the index date
* Had > 1 OAC prescription in the patient's medical records on the index date

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients' medical charts with newly initiating warfarin or apixaban within the identification period fulfilling the study eligibility criteria
Sampling Method: Probability Sample
Enrollment: 12354 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Incidence of major bleeding among oral anticoagulant (OAC) initiators | Maximum 3 years

SECONDARY OUTCOMES:
Incidence of thromboembolic events | Maximum 3 years
Incidence of stoke/SE (secondary event) among OAC initiators | Maximum 3 years
Incidence of major bleeding and stoke/SE (secondary event) among OAC initiators stratified by CCr | Maximum 3 years
  CCr creatinine clearance (< 50ml/min and > 50ml/min)
Incidence of cardiovascular/all cause death among OAC initiators | Maximum 3 years
Incidence of myocardial infarction among OAC initiators | Maximum 3 years
Incidence of major adverse cardiac event among OAC initiators | Maximum 3 years
Incidence of cardiovascular/all cause death among OAC initiators stratified by CCr (creatinine clearance rate) | Maximum 3 years
  CCr (< 50ml/min and > 50ml/min)
Incidence of myocardial infarction among OAC initiators stratified by CCr | Maximum 3 years
  CCr (< 50ml/min and > 50ml/min)
Incidence of major adverse cardiac event among OAC initiators stratified by CCr | Maximum 3 years
  CCr (< 50ml/min and > 50ml/min)
Distribution of clinical characteristics among OAC initiators | Maximum 3 years
  Clinical characteristics will be summarized using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Minato-ku, Tokyo, Japan

REFERENCES:
- [Derived] Morimoto T, Hoshino H, Matsuo Y, Ibuki T, Miyata K, Koretsune Y. Safety and Effectiveness of Apixaban Versus Warfarin in Japanese Patients with Nonvalvular Atrial Fibrillation Stratified by Renal Function: A Retrospective Cohort Study. Am J Cardiovasc Drugs. 2023 Nov;23(6):721-733. doi: 10.1007/s40256-023-00611-7. Epub 2023 Oct 17. PMID 37847442
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm